CLINICAL TRIAL: NCT00276627
Title: Enhancing Patient-Oncologist Communication
Brief Title: Computer Program in Improving Communication Between Doctors and Patients With Stage IV Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00010216; DUMC-4510-05-2RER; CDR0000452788 (Other: NCI)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — CD-ROM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- communication lecture (Active Comparator)
  Interventions: Behavioral: communication lecture
- lecture plus CD-ROM (Experimental)
  Interventions: Behavioral: lecture plus CD-ROM

INTERVENTIONS:
Behavioral: communication lecture — lecture on communication skills with oncology patients
  Arms: communication lecture
Behavioral: lecture plus CD-ROM — Interactive CD-ROM about responding to patients' negative emotions. The CD-ROM included tailored feedback on the oncologists' own recorded conversations.
  Arms: lecture plus CD-ROM

SUMMARY:
RATIONALE: A computer program and education materials may help improve the ability of doctors to communicate with patients.

PURPOSE: This randomized clinical trial is studying how well a computer program together with education materials works in improving communication between doctors and patients with stage IV cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the impact of a CD-ROM-based intervention in improving communication behaviors between oncologists and patients with stage IV cancer.
* Compare the quality of audio-recorded conversations between oncologists and patients with advanced cancer with best practices described in the literature, with particular attention to communication behaviors that promote patient disclosure of concerns, use of emotion handling skills, recognition of empathic opportunities, and the conveying of prognostic information and compare.
* Develop an intervention to improve oncologists' communication skills in these areas using an interactive CD-ROM based on the oncologists' own recorded discussions with patients.
* Determine the feasibility of this intervention and, using a randomized, controlled design, measure its effectiveness for changing physician communication behaviors and relevant patient outcomes including reduced distress and increased satisfaction.

OUTLINE: This is a randomized, controlled, 3-part, multicenter study.

* Part 1 (baseline): Patients undergo an audio-recorded outpatient encounter with their oncologist to see how oncologists elicit patients' concerns and respond to emotional content. Within 1 week later, patients undergo a 10-minute interview by telephone.
* Part 2 (intervention): Oncologists are randomized to 1 of 2 arms.

  * Arm I (intervention): Oncologists receive a personalized, user-friendly CD-ROM that contains their coded conversations, packaged with related educational material to be used for 3 months.
  * Arm II (control): Oncologists do not receive a CD-ROM or any other educational material support.
* Part 3 (post-intervention): Three months later, oncologists in both arms are reassessed by recording another 400 clinic visits between the same oncologists and a new group of patients to measure the intervention impact.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced cancer (stage IV disease) AND meets all of the following criteria:

  * Referred by participating physician
  * Must speak English
  * Receiving primary oncology care at participating centers, defined as at least 2 visits to the clinic during the past year and a future scheduled appointment
  * Receiving treatment for any malignancy
  * Has access to a telephone

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2003-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of empathic statements and responses to patients' expressions of negative emotion | Postintervention audio recordings and follow-up surveys
  Postintervention audio recordings were used to identify the number of empathic statements and responses to patients' expressions of negative emotion. Surveys evaluated patients' trust in their oncologists and perceptions of their oncologists' communication skills.

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tulsky, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Cancer Institute, Durham, North Carolina
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Tulsky JA, Arnold RM, Alexander SC, Olsen MK, Jeffreys AS, Rodriguez KL, Skinner CS, Farrell D, Abernethy AP, Pollak KI. Enhancing communication between oncologists and patients with a computer-based training program: a randomized trial. Ann Intern Med. 2011 Nov 1;155(9):593-601. doi: 10.7326/0003-4819-155-9-201111010-00007. PMID 22041948